CLINICAL TRIAL: NCT05137548
Title: A Phase 1, Open-label, 2-cohort, Multiple Dose, Drug-drug Interaction, Safety and Tolerability, Fixed-sequence Study to Investigate the Potential Interaction Between ATI-2173 When Coadministered With Tenofovir Disoproxil Fumarate in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study Between ATI-2173 and Tenofovir Disoproxil Fumarate in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antios Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANTT102
Record Dates: First submitted 2021-10-27; First posted 2021-11-30 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Tenofovir; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATI-2173. (Experimental): ATI-2173
  Interventions: Drug: ATI-2173 50 mg
- Tenofovir Disoproxil Fumarate (Experimental): Tenofovir disoproxil fumarate
  Interventions: Drug: Tenofovir 300Mg Oral Tablet

INTERVENTIONS:
Drug: ATI-2173 50 mg — ATI-2173 is a liver-targeted phosphoramidate oral prodrug of clevudine designed to enhance anti-HBV activity while decreasing systemic exposure to clevudine. It will be dosed as a capsule by mouth
  Arms: ATI-2173.
Drug: Tenofovir 300Mg Oral Tablet — Tenofovir is an oral nucleotide analogue reverse transcriptase inhibitor used for chronic hepatitis B virus. It will be dosed as a tablet by mouth
  Other Names: Viread 300 mg
  Arms: Tenofovir Disoproxil Fumarate

SUMMARY:
This study is a single-center, open-label, 2-cohort, multiple dose, fixed-sequence, DDI study in healthy adult subjects. Healthy volunteers will be administered multiple oral doses of ATI-2173 in combination with tenofovir disoproxil fumarate and assessed for safety and tolerability including blood tests to show how the body metabolizes and eliminates the investigational drug as well as how the investigational drug interacts with tenofovir disoproxil fumarate.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated Informed Consent Form (ICF)
2. Stated willingness to comply with all study procedures (including ability and willingness to abstain from alcohol from 48 hours prior to the first study drug administration until discharge) and availability for the duration of the study
3. Healthy adult male or female
4. Aged between 18 and 59 years, inclusive
5. Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
6. Non- or ex-smoker (an ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
7. Suitable veins for cannulation or repeated venipuncture as assessed by an Investigator at Screening Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an Investigator

9. Agrees to abstain from blood or plasma donation from the Screening visit until 3 months after the last study drug administration 10. If female, must meet one of the following criteria:

1. Is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include:

   * Abstinence from heterosexual intercourse from Screening through to at least 60 days after the last dose of the study drug
   * Male partner vasectomized at least 180 days prior to Screening
   * Double-barrier method (eg, male condom, spermicide and diaphragm or cervical cap used simultaneously) from Screening through to at least 30 days after the last dose of the study drug
   * One of the following contraceptive methods with a barrier method (eg, male condom) from at least 28 days prior to the first study drug administration through to at least 60 days after the last dose of the study drug:
   * Systemic contraceptives (combined birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
   * Intrauterine device (with or without hormones) If systemic contraceptives are used, must agree to use an additional acceptable non-hormonal method during the study and for at least 60 days after the last dose of the study drug Or
2. Is of non-childbearing potential, defined as surgically sterile (ie, has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a postmenopausal state (at least 1 year without menses without an alternative medical condition prior to Screening), as confirmed by follicle-stimulating hormone levels (≥ 40 mIU/mL).

   11. A male study subject that engages in sexual activity that has the risk of pregnancy must:
   * Agree to use a double-barrier method (eg, male condom, spermicide and diaphragm or cervical cap used simultaneously) or be abstinent from heterosexual intercourse from Screening to at least 90 days after the last study drug administration or be unable to procreate; defined as surgically sterile (i.e. has undergone a vasectomy at least 180 days prior to Screening) AND
   * Agree to not donate sperm during the study and for at least 90 days after the last study drug administration 12. Body weight ≥35 kg (≥77 lb)

   Exclusion Criteria:
   1. Female who is lactating
   2. Female who is pregnant according to the pregnancy test at Screening or prior to the first study drug administration
   3. Pulse rate less than 50 beats per minute or more than 100 beats per minute at Screening or prior to the first study drug administration unless deemed not clinically significant by the Investigator
   4. Blood pressure below 100/60 mmHg or higher than 140/90 mmHg at Screening or prior to the first study drug administration unless deemed not clinically significant by the Investigator
   5. History of hypersensitivity to ATI-2173, clevudine, tenofovir, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
   6. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability including but not limited to cholecystectomy
   7. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease, in the opinion of an Investigator
   8. Presence of clinically significant ECG abnormalities at Screening or prior to study drug administration, in the opinion of an Investigator
   9. Presence of clinically significant muscle disorders, myopathies or other forms of liver disease, in the opinion of an Investigator
   10. Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m2 using the Modification of Diet in Renal Disease (MDRD) equation at Screening or < 60 mL/min/1.73 m2 on Day -1
   11. Hemoglobin value below the lower limit of the reference laboratory at Screening or prior to study drug administration
   12. Unexplained persistent elevations of serum transaminases or creatine kinase (CK) levels at Screening or prior to study drug administration
   13. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
   14. Any clinically significant illness in the 28 days prior to the first study drug administration
   15. Use of any prescription drugs (except systemic contraception and intrauterine devices) in the 30 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy
   16. Use of St. John's wort in the 30 days prior to the first study drug administration
   17. Use of quinine-containing products (eg, tonic water), grapefruit products, pomelo products, Seville orange products, including supplements containing Citrus aurantium or "bitter orange", in the 14 days prior to the first study drug administration
   18. Any history of latent or active tuberculosis
   19. Positive screening tuberculosis blood test
   20. Immunization with a COVID-19 vaccine in the 14 days prior to the first study drug administration
   21. Scheduled immunization with a COVID-19 vaccine (first or second dose) during the study that, in the opinion of an investigator, could potentially interfere with subject participation, subject safety, study results, or any other reason
   22. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first drug administration
   23. Positive test results for HIV-1/HIV-2 antibodies, hepatitis B surface antigen or hepatitis C antibody at Screening
   24. Any other clinically significant abnormalities in laboratory test results at Screening or prior to the first drug administration that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
   25. Inclusion in a previous group for this clinical study
   26. Participation in another clinical study with a non-biologic Investigational Product (IP) or new formulation of a marketed non-biologic drug in the 30 days prior to the first study drug administration
   27. Participation in another clinical study with a biologic (marketed or investigational) in the 90 days or 5 half-lives (whichever is longer) prior to the first study drug administration
   28. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
   29. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration
   30. History of pathologic fracture or other risk factors for osteoporosis or bone loss

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Cmax of ATI-2173, clevudine, and M1 in plasma | Through end of study, approximately 3 months
AUCtau of ATI-2173, clevudine, and M1 in plasma | Through end of study, approximately 3 months
AUC0-t of ATI-2173, clevudine, and M1 in plasma | Through end of study, approximately 3 months
Cmax of tenofovir | Through end of study, approximately 3 months
Cmin,ss of tenofovir | Through end of study, approximately 3 months
AUC0-tau of tenofovir | Through end of study, approximately 3 months
AUC0-t of tenofovir | Through end of study, approximately 3 months

SECONDARY OUTCOMES:
Number of Adverse Events | Through end of study, approximately 3 months

OTHER OUTCOMES:
Plasma trough concentrations of tenofovir, ATI-2173, clevudine, and M1 | Days 18, 19, 20 and 21

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No